CLINICAL TRIAL: NCT00847028
Title: Oral Glucose Solution as Pain Relief in Newborns: Results of a Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Prof. Monique M. Elseviers, Nusing Sciences, University of Antwerp
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HHmol-001; (EC NR 7/37/203).
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Pain
Keywords: Newborn; Pain; glucose solution; venipuncture; non-pharmacologic pain relief.
MeSH Terms: conditions — Pain | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): glucose 10%
  Interventions: Other: glucose 10%
- 2 (Experimental): glucose 20%
  Interventions: Other: 20% glucose
- 3 (Experimental): glucose 30%
  Interventions: Other: glucose 30%
- 4 (Placebo Comparator): placebo: sterile water
  Interventions: Other: sterile water

INTERVENTIONS:
Other: glucose 10% — 2 minutes prior to the venipuncture, a 10% glucose concentration was administered orally
  Arms: 1
Other: 20% glucose — 2 minutes prior to the venipuncture, a 20% glucose concentration was administered orally
  Arms: 2
Other: glucose 30% — 2 minutes prior to the venipuncture, a 30% glucose concentration was administered orally
  Arms: 3
Other: sterile water — 2 minutes prior to the venipuncture, sterile water was administered orally
  Arms: 4

SUMMARY:
This study investigates which concentration of glucose is most effective in reducing pain for venipuncture in the newborn.

DETAILED DESCRIPTION:
This double-blind clinical trial is conducted on a maternity and newborn (N*) ward. Each time, during at least one month, one of the four selected solutions (glucose 10%, 20%, 30% and placebo) will be administered orally, 2 minutes prior to the venipuncture. The pain from the skin puncture will be scored using a validated pain scale (the "Leuven" pain scale).

ELIGIBILITY:
Inclusion criteria

* Neonates were included if they had to undergo a venipuncture as part of routine medical care.

Exclusion criteria

* Unstable neonates with respiratory support as well as neonates with a proven neurological abnormality were excluded.
* Newborns who had been administered sedatives, analgesics or naloxone during the past 48 hours were excluded along with premature infants younger than 32 weeks post menstrual age.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Pain after venipuncture measured by the Leuven pain scale for newborns | solution administration- waiting for 2 minutes-then venipuncture and immediate pain scoring

SECONDARY OUTCOMES:
difference in heart rhythm | heart rhythm measured before painful procedure - heart rythm after venipuncture compared to baseline measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ben Dilen, MSN, Principal Investigator — Universiteit Antwerpen + Heilig Hart ziekenhuis Mol
Locations (1):
- H Hart ziekenhuis, Mol, Antwerp, Belgium